CLINICAL TRIAL: NCT05851157
Title: A Phase 1, Randomized, Open-label, Crossover Study Evaluating the Effects of Food on the Pharmacokinetics of VX-548 in Healthy Adults
Brief Title: A Study to Evaluate the Effect of Food on the Pharmacokinetics of VX-548
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX22-548-016
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-548 (Experimental): Participants will be randomized to receive a single dose of VX-548 in 1 of 6 treatment sequences with 3 dosing periods to assess different fed conditions and timing of meal administration on the PK of VX 548. There will be a 14 day washout period between each dosing period.
  Interventions: Drug: VX-548

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety, and tolerability of VX-548 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 35.0 kilogram per meter square (Kg/m^2)
* A total body weight greater than (>) 50 kilogram (kg)

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* Participants of childbearing potential

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-548 and its Metabolite | Pre-dose up to Day 35 Post-dose
Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-tlast) of VX-548 and its Metabolite | Pre-dose up to Day 35 Post-dose
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-548 and its Metabolite | Pre-dose up to Day 35 Post-dose

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 44

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing